CLINICAL TRIAL: NCT05492019
Title: Effect of Doxycycline in Levodopa Treated Parkinson's Disease Patients: Randomized, Double-Blind, Placebo-Controlled Trial.
Brief Title: Effect of Doxycycline in Levodopa Treated Parkinson's Disease Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr. Shahanaz Parvin, MBBS, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3914
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Parkinson Disease
Keywords: "Parkinson's disease" "Doxycycline"
MeSH Terms: conditions — Parkinson Disease | interventions — Doxycycline

STUDY DESIGN:
Intervention Model Description: The patients will be randomly allocated into two arms: control and intervention. Patients in intervention arm consisted of 30 patients who will receive levodopa plus doxycycline orally for 8 weeks. On the other hand, control arm consisted of 30 patients who will receive levodopa plus placebo for 8 weeks.
Who Masked: Participant, Investigator
Masking Description: Participants and investigators will not know which arm patients have been assigned to or if they receive doxycycline or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doxycyline- Patients receiving Doxycycline . (Experimental): Drug generic name: Doxycycline Dosage form- oral capsule Dosage- (50mg) one capsule Frequency- twice daily Duration- 8 weeks.
  Interventions: Drug: Doxycycline
- Control- Patients receiving placebo (Placebo Comparator): Patient will receive one capsule of placebo twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Doxycycline — Doxycycline 50 mg capsule twice daily for 8 weeks.
  Other Names: Brand name- Doxin
  Arms: Doxycyline- Patients receiving Doxycycline .
Drug: Placebo — Oral placebo identical to Doxycycline
  Arms: Control- Patients receiving placebo

SUMMARY:
This study is a Randomized, Double-Blind, Placebo-Controlled Trial. The objective of the study is to assess the effect of doxycycline in levodopa treated Parkinson's disease patients regarding motor performance and cognitive functions. Parkinson's disease patients on levodopa medications will be assigned to receive doxycycline 50mg twice daily or placebo over 8 weeks. The motor and cognitive symptoms of Parkinson's disease will be assessed after 4 weeks and 8 weeks follow up.

DETAILED DESCRIPTION:
Parkinson's disease is a progressive neurodegenerative disorder that is caused by degeneration of dopaminergic neuron in the substantia nigra. Most commonly used drug, levodopa can improve the dopamine level in brain but cannot give neuroprotection and also induces motor fluctuations and dyskinesia in many patients. Doxycycline has been shown anti-inflammatory and neuroprotective effects against Parkinson's disease on animal model. It also reduced Levodopa induced dyskinesia without compromising the motor benefits of Levodopa. Therefore, the present study is to attempt to improve the sign symptoms of Parkinson's disease by giving doxycycline along with Levodopa.

This study is a Randomized, Double-Blind, Placebo-Controlled Trial and conducting at Department of Pharmacology, BSMMU in collaboration with Department of Neurology, BSMMU. A total of 60 patients suffering from Parkinson's disease is selected according to inclusion and exclusion criteria. The diagnosis of the patients suffering from Parkinson's disease will be performed by a neurologist at movement disorder clinic of department of Neurology, BSMMU. Patients will undergo MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) to assess the severity of the disease. The patients will be randomly allocated into two arms: control and intervention. Patients in intervention arm consisted of 30 patients who will receive levodopa plus doxycycline orally for 8 weeks. On the other hand, control arm consisted of 30 patients who will receive levodopa plus placebo for 8 weeks. The severity of Parkinson's disease will be assessed after 4 weeks and 8 weeks follow up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Parkinson's disease patient taking Levodopa
* Age: More than 18 years
* Sex: All

Exclusion Criteria:

* Secondary causes of parkinsonism
* Atypical parkinsonian syndromes
* Prior stereotaxic surgery for Parkinson's disease
* Known hypersensitivity to doxycycline
* Pregnancy and lactation
* Suffering from active malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Effect of doxycycline on improvement of motor performance and cognitive functions of Parkinson's disease. | 8 weeks
  Assessing and comparing the severity of symptoms of Parkinson's disease of two groups by using MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) at baseline, 4 weeks and 8 weeks following doxycycline and placebo supplementation.

SECONDARY OUTCOMES:
High sensitive C-reactive protein | 8 weeks
  will be measured before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Shahanaz Parvin, MBBS, Principal Investigator — Bangabandhu Sheikh Mujib Medical University (BSMMU)
Locations (1):
- Bangabandhu Sheikh Mujib Medical University (BSMMU), Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No